CLINICAL TRIAL: NCT03164798
Title: Serum BDNF Role as a Biomarker for Stroke Rehabilitation
Acronym: BDNF
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Hyuk Chang, Associate Professor, Samsung Medical Center
Other Study IDs: 2016-08-059
Record Dates: First submitted 2017-05-21; First posted 2017-05-24 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Biomarker; Rehabilitation; BDNF
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BDNF Val66Met polymorphism
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Conventional inpatient rehabilitation — comprehensive inpatient rehabilitation for 2 weeks

SUMMARY:
This study aims to develop the quantitative biomarker to establish the individualized strategy in stroke rehabilitation. Brain-derived neurotrophic factor (BDNF) acts on certain neurons of the central nervous system (CNS) helping to support the survival of existing neurons, and encourage the growth and differentiation of new neurons and synapses. BDNF in CNS can be assessed by analysing serum BDNF. The final objective of this study is to demonstrate a role of biomarker of BDNF in stroke rehabilitation to establish the individualized strategy.

DETAILED DESCRIPTION:
Serum BDNF, proBDNF and MMP-9 in all participants will be measured before and after the comprehensive inpatient rehabilitation during subacute stroke phase. At 3 months after stroke onset, serum BDNF, proBDNF and MMP-9 will also be measured.

In addition, motor impairment with Fugl-Meyer assessement will be assessed at same time points with serum analysis.

We will compare potential serum biomarkers with motor impairment in stroke patients

ELIGIBILITY:
Inclusion Criteria:

* unilateral stroke patients
* admission to the rehabilitation department before 1 month after stroke onset
* mild to severe motor impairment at time of transferring to the rehabilitation department

Exclusion Criteria:

* Progressive or unstable stroke
* Pre-existing and active major neurological disease
* Pre-existing and active major psychiatric disease
* Advanced liver, kidney, cardiac, or pulmonary disease
* A terminal medical diagnosis consistent with survival < 1 year)
* Pregnant or lactating woman

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subacute stroke patients who were received the comprehensive inpatients rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Serum BDNF | At 2 weeks after the comprehensive inpatient rehabilitation
  serum BDNF level

SECONDARY OUTCOMES:
Serum proBDNF | At 2 weeks after the comprehensive inpatient rehabilitation
  Serum proBDNF level
MMP-9 | At 2 weeks after the comprehensive inpatient rehabilitation
  MMP-9 level

CONTACTS AND LOCATIONS:
Overall Officials: Won Hyuk Chang, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Chang WH, Bang OY, Shin YI, Lee A, Pascual-Leone A, Kim YH. BDNF polymorphism and differential rTMS effects on motor recovery of stroke patients. Brain Stimul. 2014 Jul-Aug;7(4):553-8. doi: 10.1016/j.brs.2014.03.008. Epub 2014 Mar 26. PMID 24767962
- [Background] Hwang JM, Kim YH, Yoon KJ, Uhm KE, Chang WH. Different responses to facilitatory rTMS according to BDNF genotype. Clin Neurophysiol. 2015 Jul;126(7):1348-53. doi: 10.1016/j.clinph.2014.09.028. Epub 2014 Oct 12. PMID 25454277
- [Background] Uhm KE, Kim YH, Yoon KJ, Hwang JM, Chang WH. BDNF genotype influence the efficacy of rTMS in stroke patients. Neurosci Lett. 2015 May 6;594:117-21. doi: 10.1016/j.neulet.2015.03.053. Epub 2015 Mar 26. PMID 25817361
- [Background] Chang WH, Hwang JM, Uhm KE, Pascual-Leone A, Kim YH. Corticospinal excitability in the non-dominant hand is affected by BDNF genotype. Neurol Sci. 2017 Feb;38(2):241-247. doi: 10.1007/s10072-016-2749-9. Epub 2016 Oct 25. PMID 27783184